CLINICAL TRIAL: NCT02906280
Title: Randomized Controlled Trial Comparing the Performance of 19 Gauge Versus 22 Gauge EBUS-TBNA Needles in Lung Carcinoma
Brief Title: RCT Comparing 19Ga vs 22Ga EBUS-TBNA Needles in Carcinoma.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Christophe Dooms, MD, PhD, MD, PhD, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S58667
Record Dates: First submitted 2016-05-27; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Lung Neoplasm
Keywords: EBUS-TBNA
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 19 Ga EBUS-TBNA needle (Experimental): needle aspiration by a flexible 19 Ga needle (Olympus)
  Interventions: Device: EBUS-TBNA needle
- 22 Ga EBUS-TBNA needle (Active Comparator): needle aspiration by a 22 Ga needle (Olympus)
  Interventions: Device: EBUS-TBNA needle

INTERVENTIONS:
Device: EBUS-TBNA needle — tissue sampling

SUMMARY:
EBUS-TBNA is often the sole diagnostic test applied in patients with stage IV lung cancer. A limitation of the TBNA needle when using a 22 Gauge needle is the limited ability to procure adequate histological samples. Although a larger 19 Ga needle can procure histological samples as demonstrated by the conventional 19 Ga needle, published data are not existing with respect to molecular diagnostics. A new nitinol-based 19 Ga needle has been developed for EBUS-TBNA. Given the frequent usage of 22 Ga needles for molecular diagnostics and the recent technical advancements in 19 Ga needle technology, we conduct a RCT to compare the performance of both needle types.

DETAILED DESCRIPTION:
All patients with (suspected) stage IV lung carcinoma identified on spiral computed tomography scan and requiring an EBUS-TBNA investigation to obtain intrathoracic hilar or mediastinal lymph node tissue for diagnosis, subtyping and genotyping of lung cancer are eligible for participation in this study. Procedural technique : patients undergo an EBUS-TBNA procedure with either the Flex 19 Ga needle or the 22 Ga needle ; all procedures are performed using a linear array echoendosope under moderate sedation (standard practice). Primary endpoint of the study is the presence of core tissue that is defined as a continuous string of material as observed on the microscopic examination. Secondary endpoints are elements relevant to molecular analysis.

ELIGIBILITY:
Inclusion Criteria:

* (suspected) stage IV lung carcinoma identified on spiral computed tomography scan
* requiring an EBUS-TBNA investigation to obtain intrathoracic hilar or mediastinal lymph node tissue for diagnosis

Exclusion Criteria:

* uncontrolled coagulopathy
* tracheal stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Tissue core | 14 months
  Descriptive tissue characteristics of tumor sample

SECONDARY OUTCOMES:
Tumor cellularity per area of diagnostic tissue | 14 months
  Objective pathologic measurement of tumor density
Quantity of DNA extracted | 14 months
  Objective measurement of the amount of DNA
Success rate of Next Generation Sequencing | 14 months
  Feasibility of NGS testing

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No